CLINICAL TRIAL: NCT06568510
Title: Coiling of Echogenic Perineural Catheters.
Brief Title: Coiling of Echogenic Sciatic Nerve Perineurial Catheters with Integral Stylet
Status: Completed | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, THEODOSIOS SARANTEAS, PROFESSOR, Attikon Hospital
Other Study IDs: 342 (date:9/05/2024)
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Pain; Trauma
Keywords: Prineural catheter; Ultrasound; Sciatic nerve
MeSH Terms: conditions — Pain; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with continuous sciatic nerve block: Patients were placed in the lateral position (with the injured leg uppermost) and a US-guided sciatic nerve block was performed under aseptic conditions . The sciatic nerve was visualized at the upper third of the posterior thigh (short axis view) and a Tuohy needle (21 G × 10 mm, was inserted in a lateral to medial direction. The needle was placed underneath the sciatic nerve and 10 ml of ropivacaine (0.1%) were injected. A perineural catheter (with retracted integral stylet by 6 cm) was then threaded through the needle tip and coiled behind the sciatic nerve. Confirmation of correct catheter tip placement was defined as adequate spread and contact of ropivacaine injectate (3 ml, 0.1%) with the sciatic nerve
  Interventions: Procedure: Continuous peripheral nerve block

INTERVENTIONS:
Procedure: Continuous peripheral nerve block — A perineurial catheter is placed to a nerve structure through a Touchy needle

SUMMARY:
Coiling of perineurial catheters under the sciatic nerve and examination of catheters position through ultrasound imaging 36 hours postoperatively.

DETAILED DESCRIPTION:
To assess procedural effectiveness of the preferred coiling technique (method B), a pilot study was performed. Straight perineural catheters with coiled distal ends behind the sciatic nerve were examined in 25 patients who had sustained tibia fractures.

Patients were placed in the lateral position (with the injured leg uppermost) and a US-guided sciatic nerve block was performed under aseptic conditions. The sciatic nerve was visualized at the upper third of the posterior thigh (short axis view) and a Tuohy needle (21 G × 10 mm, SonoLong/NanoLine, PAJUNK, Germany) was inserted in a lateral to medial direction. The needle was placed underneath the sciatic nerve and 10 ml of ropivacaine (0.1%) were injected. A perineural catheter (with retracted integral stylet by 6 cm) (SonoLong Sono, PAJUNK, Germany) was then threaded through the needle tip and coiled behind the sciatic nerve. Confirmation of correct catheter tip placement was defined as adequate spread and contact of ropivacaine injectate (3 ml, 0.1%) with the sciatic nerve (Figure 2C). If the distribution of the local anaesthetic (LA) could not be visualized on the first infusion, 2 additional injections were performed until the distribution was clearly seen. If LA spread could not be visually confirmed, or if, when confirmed, LA did not come in contact with the sciatic nerve, the case was excluded.

Subcutaneous tunneling (4 cm long) and placement of a transparent adhesive dressing were used to secure the catheter. All sciatic nerve blocks were followed by an adductor canal block (10 ml of ropivacaine 0.5%) and general anaesthesia. A continuous infusion of ropivacaine (8-12 ml, 0.1%) was commenced and a combination of oxycodone 5 mg with paracetamol 325 mg was provided on an as-needed basis after surgery.

All nerve blocks were assessed and data were collected in the post-anaesthetic care unit, and every 12 hours thereafter until 36 hours postoperatively from members of acute pain service (APS) team not participating in the study.

ELIGIBILITY:
Inclusion Criteria: Orthopaedic patients with Tibia fractures

-

Exclusion Criteria:

* Patients with infection in the sub gluteal region.
* Allergies to local aesthetics
* Patients refusal to consent for the nerve block
* Neurological disorders
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopaedic patients with Tibial fractures
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Rate of correct placement of coiled perineural catheters under the sciatic nerve | 10 minutes
  A Tuohy needle is placed underneath the sciatic nerve. Then, a catheter is headed out through the curved tip of the Tuohy needle and coils underneath the sciatic nerve. Catheter's position was assessed after 36 hour postoperatively. Catheters tip internal displacement was assessed after contact with the nerve of 3 cc of local anesthetic injecting via the catheter (maximum three tines).

CONTACTS AND LOCATIONS:
Overall Officials: Mavrogenis Andreas, Principal Investigator — Academic teacher
Locations (1):
- Department of anesthesia ,ATTIKON UNIVERSITY HOSPITAL OF ATHENS, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saranteas T, Poulogiannopoulou E, Ntalamagka G, Skaligkou P, Giasafaki M, Papadimos T. Perineural coiled echogenic catheters with a flexible distal end: A brief technical report. Anaesth Crit Care Pain Med. 2024 Apr;43(2):101341. doi: 10.1016/j.accpm.2023.101341. Epub 2023 Dec 22. No abstract available. PMID 38142867
- [Derived] Saranteas T, Poulogiannopoulou E, Riga M, Panagouli K, Mavrogenis A, Papadimos T. Coiling of echogenic perineural catheters with integral stylet: A proof-of-concept randomized control trial in a sciatic nerve block simulator and a pilot study in orthopaedic-trauma patients. F1000Res. 2024 Dec 2;13:1103. doi: 10.12688/f1000research.155381.2. eCollection 2024. PMID 39639915
- See also: doi — https://doi.org/10.1016/j.accpm.2023.101341